CLINICAL TRIAL: NCT00656552
Title: Safety and Efficacy of Escitalopram in the Treatment of Premature Ejaculation A Double-Blind, Placebo-Controlled, Fixed-Dose,Randomized Controlled Study
Brief Title: Safety and Efficacy of Escitalopram in the Treatment of Premature Ejaculation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: kasr elainy school of medicine, Gamal Soltan
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EPE100
Record Dates: First submitted 2008-04-07; First posted 2008-04-11 (Estimated); Last update posted 2008-04-11 (Estimated); Status verified 2008-04

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Escitalopram — Patient undergo a double- blind therapy of Escitalopram (10 mg) orally daily during breakfast (n=50) or placebo (n=50) for four weeks.

SUMMARY:
Escitalopram has been claimed to have the highest selectivity for the human serotonin transporter relative to the noradrenaline or dopamine transporters. This might be associated with greater clinical efficacy. Most adverse events reported by escitalopram-treated patients are mild and transient.

In this study, we compare escitalopram with placebo in the treatment of PE.

DETAILED DESCRIPTION:
Safety and Efficacy of Escitalopram in the Treatment of Premature Ejaculation A Double-Blind, Placebo-Controlled, Fixed-Dose, Randomized controlled Study

Introduction

From an epidemiological perspective, premature ejaculation (PE) has been reported as the most common male sexual dysfunction with overall prevalence rates estimated at around 30% .(Laumann et al., 1999).

PE is defined by the Diagnostic and Statistical Manual of Mental Disorders(revision IV) (DSM-IV-TR) as 'the persistent or recurrent ejaculation with minimal stimulation before, on, or shortly after penetration and before the person wishes it'. (American Psychiatric Association, 1994).

ISSM Definition of Premature Ejaculation is a male sexual dysfunction characterized by ejaculation which always or nearly always occurs prior to or within about one minute of vaginal penetration; and inability to delay ejaculation on all or nearly all vaginal penetrations; and negative personal consequences, such as distress, bother, frustration and/or the avoidance of sexual intimacy (www.issm.info).

Premature ejaculation has been associated with erosion in sexual self-confidence and low sexual satisfaction in men and their female partners.( Byers & Grenier ; 2003).

Behavioral therapy and psychological counseling are the historically initial approaches in the treatment of PE.However There is no evidence that non-drug therapy is able to guarantee long-term cure or improvement of PE. (Rosen, 2004).

These techniques require active involvement of the patients and their partners and the benefits are generally short-lived, and patients usually relapse. In addition, these therapies may not be applicable for some cultural and socioeconomic groups. Therefore, some pharmacological agents have been proposed for the treatment of PE(Rosen, 2004).

The serotoninergic system has an inhibitory effect on the ejaculatory reflex. Selective serotonin reuptake inhibitors (SSRIs) (paroxetine, fluoxetine, sertraline, citalopram) are reported to be effective for treating PE (Rosen, 2004; Safarinejad & Hosseini, 2006). Psychopharmacological studies suggest that PE might be due to decreased serotonergic neurotransmission through pathways that control ejaculation (Waldinger et al., 1998).

Ejaculation delay induced by SSRIs is due to alterations in specific serotonin receptors in the central nervous system. The ejaculation-retarding effect of 5-hydroxytryptamine (5-HT, serotonin) has been attributed to the activation of 5-HT1B and 5-HT2C receptors. By contrast, stimulation of 5-HT1A receptors has a facilitator effect on ejaculation (Giuliano, 2007). The net effect of acute SSRI administration is only a mild increase of 5-HT neurotransmission and mild stimulation of the various post-synaptic serotonin receptors (Waldinger et al., 2005). In contrast, chronic SSRI administration is associated with more 5-HT (serotonin) release into the synapse, stronger increase of 5-HT neurotransmission, and as a result durable activation of post-synaptic 5-HT receptors (Blier et al., 1988).

Escitalopram has been claimed to have the highest selectivity for the human serotonin transporter relative to the noradrenaline or dopamine transporters.(Owens et al; 2001) This might be associated with greater clinical efficacy. Most adverse events reported by escitalopram-treated patients are mild and transient (Lepola et al; 2003).

In this study, we compare escitalopram with placebo in the treatment of PE.

Objectives:

The objective of the present trial is to assess the safety & efficacy of Escitalopram in the treatment of premature ejaculation.

Study design:

A Double-Blind, Placebo-Controlled, Fixed-Dose, Randomized Controlled Study.

Setting:

The outpatient clinic of sexual health Kasr El-Einy (Cairo University Hospital), Cairo, Egypt.

Patients:

One hundred married patients seek medical help for what they consider premature ejaculation with possible sexual intercourse equal or greater than 1 per week.

Randomization and Allocation Concealment Randomization will be performed using allocation concealment random assignment schedule for each patient. It will be accomplished using numbered cards in closed envelopes that assured an equal number of patients in the two treatment groups.

Exclusion criteria

* Erectile dysfunction accounting to Arabic version of IIEF(International Index of Erectile Dysfunction)
* Chronic psychiatric or physical illness.
* Alcohol or substance abuse.
* Use of psychotropic and antidepressant medication.
* Patient with prostatitis
* Organic illness causing limitation of SSRI use.

Methods:

Assessment of patient:

1. History taking.
2. General examination.
3. Local genital examination.
4. Self administration of IIEF (Arabic version)
5. Pretreatment IELT(Intravaginal Ejaculatory Latency Time) measured at least 3 times.

Interventions:

Patient undergo a double- blind therapy of Escitalopram (10 mg) orally daily during breakfast (n=50) or placebo (n=50) for four weeks.

Outcome measure:

Primary outcome: change in geometric mean IELT from baseline to four weeks.

Secondary outcome: changes in the intercourse satisfaction domain values of IIEF(Arabic version).

Assessment of possible side effects

ELIGIBILITY:
Inclusion Criteria:

* One hundred married patients seek medical help for what they consider premature ejaculation with possible sexual intercourse equal or greater than 1 per week.

Exclusion Criteria:

* Erectile dysfunction accounting to Arabic version of IIEF(International Index of Erectile Dysfunction)
* Chronic psychiatric or physical illness.
* Alcohol or substance abuse.
* Use of psychotropic and antidepressant medication.
* Patient with prostatitis
* Organic illness causing limitation of SSRI use.

Ages: 20 Years to 59 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
change in geometric mean IELT from baseline to four weeks. | 4 week

SECONDARY OUTCOMES:
changes in the intercourse satisfaction domain values of IIEF(Arabic version). Assessment of possible side effects | 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Hussein MH Ghanem, M D, Study Chair — Professor of Andrology & STDs
Locations (1):
- Kasr el ainy school of medicine , Cairo university, Cairo, Egypt